CLINICAL TRIAL: NCT02599818
Title: Navigation Services to Avoid Rehospitalization (NavSTAR) Among Substance Users
Brief Title: Navigation Services to Avoid Rehospitalization (NavSTAR)
Acronym: NavSTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Maryland, College Park (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-07-224; R01DA037942-01A1 (NIH)
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Opioid-use Disorder; Cocaine Use Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NavSTAR (Experimental): Participants in this arm will receive services from the NavSTAR Patient Navigation team. The Patient Navigator will work with patients for up to 3 months post-hospital discharge to resolve internal barriers (e.g., ambivalence about treatment; low motivation; competing life demands, etc.) and external barriers (e.g., lack of transportation; lack of ID card, etc.) to appropriate utilization and engagement in addiction treatment and medical care. Interventions include motivational interventions and patient navigation with proactive case management, tailored to participants' specific needs.
  Interventions: Behavioral: NavSTAR
- TAU (Treatment as Usual) (No Intervention): Participants in this arm will receive usual care, which includes in-hospital services from a multidisciplinary substance use disorder consultation liaison team.

INTERVENTIONS:
Behavioral: NavSTAR — Participants in the NavSTAR program will work with a team of case workers who will provide motivational intervention and proactive barrier resolution services using patient navigation
  Arms: NavSTAR

SUMMARY:
This study will examine the clinical effectiveness and health economic profile of services to link hospital patients with substance use disorders to addiction treatment, promote their medical stabilization, and reduce hospital re-admissions.

DETAILED DESCRIPTION:
In recent years, the problem of rehospitalization has come under intense focus as a major contributor to preventable morbidity and escalating healthcare costs. Substance use disorders are strongly associated with poor health outcomes and highly inefficient use of healthcare services, including repeat hospitalizations. Interventions that increase adherence to recommendations for outpatient medical care and substance abuse treatment could potentially help recently-hospitalized individuals with substance use disorders to avoid unnecessary rehospitalization, associated morbidity, and medical expenses. The current study is a randomized controlled trial comparing the effectiveness of Navigation Services to Avoid Rehospitalization (NavSTAR) vs. Treatment-as-Usual (TAU) for hospital patients with co-occurring medical problems and substance use disorders. Applying Andersen's theoretical model of health service utilization, NavSTAR will employ the promising strategies of Patient Navigation and motivational interventions to facilitate engagement in outpatient medical and substance abuse treatment, thereby lowering the likelihood of rehospitalization. Patient Navigators embedded within the substance abuse consultation liaison service at a large urban hospital will deliver patient-centered, proactive navigation and motivational services initiated during the hospital stay and continued for 3 months post-discharge. Participants randomized to TAU will receive usual care from the hospital and the substance abuse consultation liaison service, which includes referral to substance abuse treatment but no continued contact post-hospital discharge. Participants will be assessed at study entry and again at 3-, 6-, and 12-months follow-up on various measures of healthcare utilization, substance use, and functioning. The primary outcome of interest is time-to-rehospitalization through 12 months. In addition, a range of secondary outcomes spanning the medical and substance abuse service areas will be assessed. The study will include an economic evaluation of the cost, incremental cost-effectiveness, and cost-benefits of NavSTAR from the service provider perspective.

ELIGIBILITY:
Inclusion Criteria:

1. adult (ages 18 and older) hospital patients;
2. current DSM-5 SUD (not in remission) for alcohol, cocaine, or opioids
3. willing and able to provide informed consent.

Exclusion Criteria:

1. current enrollment in SUD treatment;
2. primary residence outside of Baltimore City;
3. pregnant;
4. terminal medical condition (e.g., planned discharge to hospice);
5. hospitalized for a suicide attempt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Time-to-Rehospitalization | 12 months
  Days to rehospitalization

SECONDARY OUTCOMES:
30-day rehospitalization rate | 30 days
  rate of rehospitalization within 30 days
Cumulative days of inpatient hospitalization | 3, 6, 12 months
  cumulative days of inpatient hospitalization
Emergency Department utilization rate | 3, 6, 12 months
  rate of Emergency Department utilization
Emergency Department visits | 3, 6, 12 months
  cumulative number of Emergency Department visits
Mortality | 3, 6, 12 months
  all-cause mortality
addiction treatment entry | 3, 6, 12 months
  rate of entry into addiction treatment
medical follow-up care | 3, 6, 12 months
  entry into recommended medical follow-up care post-hospital discharge
self-reported quality of life rating | 3, 6, 12 months
  quality of life scores as determined by the WHO-QOL BREF
alcohol use (self-report) | 3, 6, 12 months
  days of alcohol use in the past 30 days assessed via self-report
opioid use (self-report) | 3, 6, 12 months
  days of opioid use in the past 30 days assessed via self-report
cocaine use (self-report) | 3, 6, 12 months
  days of cocaine use in the past 30 days assessed via self-report
opioid use (urine test) | 3, 6, 12 months
  opioid use assessed via urine test
cocaine use (urine test) | 3, 6, 12 months
  cocaine use assessed via urine test
alcohol use disorder criteria | 3, 6, 12 months
  acute substance use disorder criteria for alcohol
opioid use disorder criteria | 3, 6, 12 months
  acute substance use disorder criteria for opioids
cocaine use disorder criteria | 3, 6, 12 months
  acute substance use disorder criteria for cocaine

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gryczynski, PhD, Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be provided upon request and execution of a data sharing agreement specific to each use request after the key analyses are completed and manuscripts have been published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After completion of key analyses and publication of planned manuscripts by the investigators.
Access Criteria: By request, contingent on approval by and execution of a data sharing agreement.

REFERENCES:
- [Derived] Nordeck CD, Kelly SM, Schwartz RP, Mitchell SG, Welsh C, O'Grady KE, Gryczynski J. Hospital admissions among patients with Comorbid Substance Use disorders: a secondary analysis of predictors from the NavSTAR Trial. Addict Sci Clin Pract. 2024 Apr 28;19(1):33. doi: 10.1186/s13722-024-00463-9. PMID 38678216
- [Derived] Mitchell SG, Monico LB, Gryczynski J, Ross T, Terplan M, O'Grady KE. Examining the Effectiveness of the FaCES Adolescent SBIRT Intervention. J Adolesc Health. 2022 Oct;71(4S):S41-S48. doi: 10.1016/j.jadohealth.2022.04.013. PMID 36122968
- [Derived] Gryczynski J, Nordeck CD, Welsh C, Mitchell SG, O'Grady KE, Schwartz RP. Preventing Hospital Readmission for Patients With Comorbid Substance Use Disorder : A Randomized Trial. Ann Intern Med. 2021 Jul;174(7):899-909. doi: 10.7326/M20-5475. Epub 2021 Apr 6. PMID 33819055